CLINICAL TRIAL: NCT05186714
Title: Mind-body Approach and Gut Microbiota in Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 122321
Record Dates: First submitted 2021-12-27; First posted 2022-01-11 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tai Chi (Active Comparator): 12 weeks of Tai Chi classes
  Interventions: Behavioral: Tai Chi versus wellness education
- Wellnes Education (Placebo Comparator): 12 weeks of Wellness Education classes
  Interventions: Behavioral: Tai Chi versus wellness education

INTERVENTIONS:
Behavioral: Tai Chi versus wellness education — 12 weeks of Tai Chi (2x/week) or a wellness education (2x/week)

SUMMARY:
This exploratory study is to compares mechanisms of mind-body exercise with wellness education program on gut microbiota for osteoarthritis as a basis for a future large-scale trial.

DETAILED DESCRIPTION:
This exploratory study is to determine the effect of mind-body exercise on gut microbiota in patients with osteoarthritis. We will randomize 80 eligible individuals who meet the American College of Rheumatology criteria for osteoarthritis into Tai Chi or wellness education interventions for 12 weeks. Using 16S rRNA amplicon sequencing of fecal DNA samples we will compare the changes in gut microbiota profiles using 16S rRNA gene amplicon sequencing, and quantity of Streptococcus species using quantitative PCR, as well as their association with clinical outcomes. This exploratory study will guide the development of theoretically informed, effective treatment for a high-risk population further enlighten us about the pathogenesis of metabolic osteoarthritis pain.This proposal will provide crucial preliminary knowledge of the mechanism underlying Tai Chi mind-body therapy for metabolic osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 55 years
* Fulfills the American College of Rheumatology Criteria for symptomatic OA
* Baseline (Month 0) WOMAC pain subscale score ≥ 40

Exclusion Criteria:

* Dementia, neurological disease, cancer, cardiovascular disease, renal disease, liver disease, or other serious medical conditions limiting ability to participate in the programs.
* Factors known or likely to impact the intestinal microbiota or known to be associated with microbial translocation: antibiotic or probiotic use within the previous 4 weeks, gastrointestinal morbidity (irritable bowel syndrome, inflammatory bowel disease, history of gastrointestinal cancer or surgical resection, or acute, severe gastrointestinal symptoms requiring medical attention), opportunistic infection, and evidence of hepatitis B or C virus infection

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Gut microbiota | From Week 0, to Week 12
  Changes in gut composition, relative abundance and diversity, and Streptococcus abundance

SECONDARY OUTCOMES:
Change in Western Ontario and McMaster University Index (WOMAC) | From Week 0 to Week 12
  WOMAC version 3.1 questionnaire (pain subscale range, 0 [no pain]-20 [extreme pain]; the stiffness subscale range, 0 [no stiffness]-8 [extreme stiffness]; function subscale range, 0 [no difficulty with daily activities]-68 [extreme difficulty].
Change in Hospital Anxiety and Depression Scale | From Week 0 to Week 12
  The Hospital Anxiety and Depression Scale (range 0-21, with higher scores indicating more severe symptoms).
Change in Body mass index | From Week 0 to Week 12
  Body mass index is measured as the weight (kg) divided by the height (m). squared
PROMIS-29 | From Week 0 to Week 12
  PROMIS-29 measure assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance).
Patient Global, 0-100 cm VAS | From Week 0 to Week 12
  Global knee pain assessment (range, 0 [no pain]-100 [extreme pain]),
PROMIS Pain Interference | From Week 0 to Week 12
  PROMIS Pain Interference score (short form 6b item short form evaluating the extent to which pain interferes with physical, emotional and social activities).
Arthritis Self-efficacy | From Week 0 to Week 12
  Arthritis Self-efficacy Scale score (SD) (Range, 1-10)

CONTACTS AND LOCATIONS:
Overall Officials: Chenchen Wang, MD, MSc, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Rheumatology, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No